CLINICAL TRIAL: NCT03977857
Title: Prediction Model Based on Computed Tomography Liver Volume for Predicting Short-term Mortality in Hepatitis B-Acute-on-Chronic Liver Failure
Brief Title: Prediction Model Based on Computed Tomography Liver Volume for the Short-term Mortality in Hepatitis B Related Acute-on-Chronic
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, He Yingli, Research Associate, First Affiliated Hospital Xi'an Jiaotong University
Other Study IDs: XJTU1AF2019LSK-2019-061
Record Dates: First submitted 2019-06-05; First posted 2019-06-06 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Acute-on-Chronic Liver Failure; Hepatitis B, Chronic
Keywords: Hepatitis B; Acute-on-Chronic liver failure; liver volume; prognostic model
MeSH Terms: conditions — Acute-On-Chronic Liver Failure; Hepatitis B, Chronic; Hepatitis B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 28-day nonsurvival or transplantation: patients who died or underwent liver transplantation within 28 days since admission
- 28-day transplantation-free survival: patients who survived without liver transplantation at 28 days since admission

SUMMARY:
HBV-related acute-on-chronic liver failure (HBV-ACLF) deteriorates rapidly with a high short-term mortality. Early identification and accurate prognostic prediction was critical to improve survival rate. This study was sought to determine the liver volumetry as predictor for short-term mortality in HBV-ACLF and develop a simpler prognostic model based on liver morphology. Liver volumetry were determined from CT at admission. Univariate and multivariate logistic regression were used to identify the optimum prognostic indicators and develop prognostic model. Additionally, receiver operating characteristic curves were analyzed to evaluate the predictive ability of the model.

DETAILED DESCRIPTION:
HBV-ACLF deteriorates rapidly with a high short-term mortality and early identification and accurate prognostic prediction may be the key to make clinical decision and improve survival rate. Liver volume, non-invasively reflects the balance of structural collapse with hepatic regeneration, predicting the prognosis of liver diseases. However, there is no idea whether the liver volume is an indicator to predict the mortality of HBV-ACLF patients. The present study evaluated the difference of liver volume between 28-day survival group and non-survivals and developed a new prognostic model based on liver volume . This study highlighted the significance of liver morphology in predicting the outcome of HBV-ACLF for the first time.

ELIGIBILITY:
Inclusion Criteria:

1. age 18-70 years, male or female.
2. Acute hepatic insult manifesting as jaundice and coagulopathy, complicated within 4 weeks by ascites, and/or encephalopathy in a patient with chronic HBV infection
3. Abdominal CT examination was performed within 3 days after admission
4. Biochemical examinations were available within 3 days before or after CT scan

Exclusion Criteria:

1. Patients with evidence of non-B hepatitis virus: alcohol abuse leads to liver failure, autoimmune leads to liver failure, oxic or other causes that might lead to liver failure
2. Past or current hepatocellular carcinoma
3. Serious diseases in other organ systems
4. Chronic liver failure
5. There was no CT imaging data or the interval between CT scan and diagnosis of liver failure >3 days

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the patients were diagnosed with hepatitis B virus-related acute-on-chronic liver failure who met with the inclusion criteria and exclusion criteria. Two cohorts of subjects were enrolled in several liver centers. In the modeling cohort, subjects were identified retrospectively from patients with acute exacerbation of chronic hepatitis B manifesting as hepatic encephalopathy (HE), upper gastrointestinal bleeding, ascites, acute jaundice and coagulopathy, referred from January 1, 2015 to December 31,2019. In the validation cohort, subjects were enrolled from external liver centers for validating the model.
Sampling Method: Probability Sample
Enrollment: 486 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Overall survival of ACLF subjects | 28 days
  Overall survival in subjects with hepatitis B virus-related acute-on-chronic liver failure will be summarized and compared with control subjects through study day 28.

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital Xi'an Jiaotong University, Xi'an, China

REFERENCES:
- [Derived] Hu C, Jiang N, Zheng J, Li C, Huang H, Li J, Li H, Gao Z, Yang N, Xi Q, Wang J, Liu Z, Rao K, Zhou H, Li T, Chen Y, Zhang Y, Yang J, Zhao Y, He Y. Liver volume based prediction model for patients with hepatitis B virus-related acute-on-chronic liver failure. J Hepatobiliary Pancreat Sci. 2022 Dec;29(12):1253-1263. doi: 10.1002/jhbp.1112. Epub 2022 Jan 25. PMID 35029044